CLINICAL TRIAL: NCT01690429
Title: Arousalanalyse Mittels Pulswellenamplitude Bei Patienten Mit Obstruktiver Schlafapnoe
Brief Title: Arousal Analysis by Pulse Wave Amplitude in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: Weinmann Geräte für Medizin GmbH + Co. KG (Industry)
Responsible Party: Principal Investigator, Karl Heinz Ruehle, Principal Investigator, Institut für Pneumologie Hagen Ambrock eV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOMNOcheck-2012
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Arousal detection; Pulse Wave Amplitude; Obstructive Sleep Apnea; Daytime sleepiness; Cardiorespiratory risk
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OSA Patients (Other)
  Interventions: Device: Somnocheck micro

INTERVENTIONS:
Device: Somnocheck micro — Study nights in sleep lab with standard polysomnography plus Somnocheck micro. The Somnocheck micro is a device with pulse oxymetry and nasal cannula, which can be worn like a wristwatch. It records information about sleep disordered breathing, oxygen saturation, and pulse wave.

SUMMARY:
Photoplethysmography is an easy non-invasive method to detect the pulse wave amplitude (PWA) from a finger. This can be measured using the Somnocheck micro system. A pulse wave amplitude decrease (PWAD) is considered to be a marker for autonomic activation. Detecting the PWAD is a surrogate marker for waking reactions (arousal) which eventually will contribute to assess sleep disruption and resulting performance deterioration. Arousal and performance deterioration and its possible improvement under continuous positive airway pressure (CPAP) therapy will be determined in this study.

DETAILED DESCRIPTION:
Patients from the sleep laboratory with verified obstructive sleep apnea syndrome (OSAS) will be asked to participate in this study.

A device is used to determine autonomic arousal over night (SOMNOcheck micro). The Somnocheck micro records oxygen saturation as well as pulse frequency and breathing, and calculates an autonomic arousal index (AAI). Somnocheck measurements will take place in two nights (baseline and with CPAP) and parallel to a standard polysomnography (PSG). The PSG provides data to analyze the arousal frequency according to ASDA rules, which will then be compared to the AAI.

Performance is determined twice (prior and after CPAP therapy) by the use of a steering simulator programme (DASS). Differences in arousal will be correlated with differences in performance (deviation from the road, reaction time). The subjects are also asked to fill out the Epworth Sleepiness Scale (ESS) twice, prior and after therapy. Aim is to compare Somnocheck and PSG measurements and daytime sleepiness with DASS and ESS.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive Sleep Apnea (AHI >5)

Exclusion Criteria:

* Suspected acute cardiac, pulmonary or neurologic disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
pulse wave amplitude (PWA) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karl Heinz Rühle, Prof. Dr., Principal Investigator — Helios Klinik Hagen
Locations (1):
- Helios Klinik Hagen, Hagen, North Rhine-Westphalia, Germany